CLINICAL TRIAL: NCT06664593
Title: Detection of Perinatal Mental Disorders
Brief Title: Screening for Depression and Anxiety in Pregnant and Postpartum Women: Evaluating Prevalence, Risk Factors, and the Stepped Screening Protocol in a Care Pathway
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 198215
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Depression, Postpartum; Puerperal Disorders; Depression During Pregnancy; Anxiety; Anxiety Disorder/Anxiety State; Stress, Psychological; Risk Factors
MeSH Terms: conditions — Depression, Postpartum; Puerperal Disorders; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 34 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- women in the perinatal period, from pregnancy until 6-8 weeks postpartum: women from pregnancy until 6-8 weeks postpartum with and without mental health problems
  Interventions: Other: integrated perinatal mental health pathway

INTERVENTIONS:
Other: integrated perinatal mental health pathway — This observational study examines whether assessing psychosocial risk factors and screening for depression and anxiety at different time points during the perinatal period, using a stepped protocol, helps to more quickly detect women with depressive and anxiety symptoms.

SUMMARY:
Having a baby is a major life event, and for some women, it can increase the risk of developing mental health issues. A recent survey in the UK found that one in five women experience mental health problems during pregnancy or after giving birth. Unfortunately, many of these problems go unnoticed without regular check-ups, and only one in ten women receive the support they need. Regular mental health screenings can help detect these problems early, ensuring women receive the right care and support.

The study at UZ Gent aims to improve how depression and anxiety are detected in pregnant and postpartum women by using a perinatal screening protocol. This protocol involves screening women for psychosocial risks around the 16th week of pregnancy, which is done by a midwife. Further screenings take place during the second trimester (around 20 weeks) and again six weeks after birth, using questionnaires to assess for depression and anxiety (Whooley, EPDS, GAD-2, GAD-7).

If the assessment of risk factors or the screening for depression and anxiety is positive, further assessment and treatment are offered at the women's clinic. A positive screening may lead to a recommendation for a diagnostic interview, such as a semi-structured interview (M.I.N.I.), with a psychiatrist, general practitioner, or psychologist to assess for possible depression or anxiety disorders. If needed, appropriate treatment will be provided.

The study will explore how common depression and anxiety are during and after pregnancy, what factors increase the risk, and whether the screening process improves early detection and treatment. The ultimate goal is to help more women get the mental health support they need during this critical time.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged ≥ 18 years, receiving regular care follow-up in a university hospital

Exclusion Criteria:

* Non-Dutch speakers were excluded. Additionally, no data were collected from women in the vulnerable care pathway, which provides psychosocial support to those facing barriers in employment, income, housing, education, and healthcare. This group includes teenage mothers (under 18), women with intellectual disabilities, new immigrants, refugees, homeless women, and those with severe psychiatric or addiction issues referred by their psychiatrist or GP.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of women receiving regular care during pregnancy and postpartum follow-up at the women's clinic of University Hospital Ghent
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
association of psychosocial and obstetric risk factors with perinatal anxiety and depression | from enrollment at 16 weeks of pregnancy to follow-up consult at 6-8 weeks postpartum
  Using a semi-structured interview, the midwife assesses psychosocial risk factors identified from a literature review. Key factors include financial and housing problems, unplanned or unwanted pregnancy, lack of social support, experiences of violence (physical, sexual, or emotional), personal and family psychiatric history, and substance use.
  Screening for depressive and anxiety symptoms followed a stepped protocol. All participants answered Yes/No to the Whooley questions (depression) and GAD-2 (anxiety). If a participant answered positively to at least one Whooley question or both GAD-2 questions, the Edinburgh Depression Scale (EDS) was administered. A score of 13 or higher on the EDS indicated a positive depression screen. If participants scored 5 or higher on the EDS-3A (anxiety subscale), the GAD-7 was administered, with a score of 15 or higher indicating a positive anxiety screen. Obstetric information was collected from the electronic patient medical records.
association between the number of (significant) risk factors and depressive and anxiety symptoms using a cumulative risk index | from enrollment at 16 weeks of pregnancy to follow-up consult at 6-8 weeks postpartum

SECONDARY OUTCOMES:
prevalence of depressive and anxiety symptoms | from enrollment at 16 weeks of pregnancy to follow-up consult at 6-8 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Lemmens, PhD, Principal Investigator — University Hospital Ghent/University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
We have decided not to share the IPD collected throughout the trial due to concerns over participant privacy and data confidentiality. Despite efforts to anonymize the data, there remains a risk that sensitive personal information could be inadvertently disclosed.

REFERENCES:
- [Background] Van Damme R, Van Parys AS, Vogels C, Roelens K, Lemmens GMD. A mental health care protocol for the screening, detection and treatment of perinatal anxiety and depressive disorders in Flanders. J Psychosom Res. 2020 Jan;128:109865. doi: 10.1016/j.jpsychores.2019.109865. Epub 2019 Nov 1. No abstract available. PMID 31838308